CLINICAL TRIAL: NCT03169595
Title: Epithelioid Hemangioma of Bone And Soft Tissue: a Benign Tumor With Metastatic Potential
Brief Title: Epithelioid Hemangioma of Bone And Soft Tissue
Acronym: EE-META
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Costantino Errani, MD, PhD., Istituto Ortopedico Rizzoli
Other Study IDs: 0033566
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Epithelioid Hemangioma of Bone; Epithelioid Hemangioma
MeSH Terms: conditions — Angiolymphoid Hyperplasia with Eosinophilia | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — Patients affected by epithelioid hemangioma treated with surgery

SUMMARY:
The controversy surrounding epithelioid hemangioma diagnosis stems from its somewhat aggressive clinical characteristics, including multifocal presentation and occasional lymph node involvement.

The investigators reviewed the clinicopathologic and radiologic characteristics of bone and soft tissue epithelioid hemangioma in patients treated at our institution with available tissue for molecular testing.

The hypothesis is that epithelioid hemangioma may present with multifocal involvement and rare loco-regional lymph node metastasis, but it remains a benign tumor with excellent prognosis.

DETAILED DESCRIPTION:
The investigators retrospectively reviewed patients treated for epithelioid hemangioma of the bone and soft tissue in a single insitution. The purpose of this study is to evaluate the pathological, clinical, and radiological characteristics of epithelioid hemangioma arising within bone and soft tissue, in the first cohort of cases where the definitive diagnosis is supplemented by molecular techniques.

The hypothesis is that the improved knowledge regarding this rare entity can more definitively elucidate the benign biology of epithelioid hemangioma.

ELIGIBILITY:
Inclusion Criteria:

* patients with epithelioid hemangioma of bone and soft tissue in the extremities and pelvis

Exclusion Criteria:

* patients with epithelioid hemangioma of bone and soft tissue in the spine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with epithelioid hemangioma of bone and soft tissue treated in a single institution
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-10-07 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Multifocal presentation of patients with epithelioid hemangioma of bone and soft tissue without producing a fatal outcome | 2 years
  The investigators defined multifocal presentation the presence of secondary lesions by imaging at presentation of the disease or during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Davide Donati, MD, Study Director — Istituto Ortopedico Rizzoli

IPD SHARING:
Plan to Share IPD: Yes
publish a manuscript in international journal